CLINICAL TRIAL: NCT06771310
Title: Effect of Kinesiotaping Versus Endurance Exercise on Postmenopausal Non Specific Low Back Pain
Brief Title: Effect of Kinesiotaping Versus Endurance Exercise on Postmenopausal Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Asmaa Mohamed Gaballah, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/002931
Record Dates: First submitted 2024-02-10; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Low Back Pain
Keywords: Kinesiotape; Endurance exercise; Postmenopausal; Low back pain.
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endurance exercise group (Experimental): The participants will perform endurance exercise (three times per week for 12 weeks
  Interventions: Other: Endurance exercise
- Kinesiotaping group (Experimental): The participants will receive kinesiotaping (replaced every five days) for 12 weeks.
  Interventions: Other: Kinesiotaping

INTERVENTIONS:
Other: Endurance exercise — The exercise-training program will be consisted of 10 minutes warming up, 30 minutes of treadmill walking, and 10 min cooling down three times per week.
  Warming up: It will be in the form of stretching of muscle groups for 10 minutes (3-5 stretch for the key muscle group (iliopsoas muscle, gluteus maximus ,quadriceps ,tibialis anterior , calf muscle, hold for 20-30 seconds), before the actual aerobic training session.
  Actual session: Participants will receive aerobic exercises in the form of Moderate aerobic exercise training in the form of 30 min of treadmill walking and corresponding to a target heart rate of 65% to 75% of HR max (Maximum HR = 220 - Age ) to be gradually achieved and maintained throughout the training program.
  Cooling down: It will be in the form of a treadmill walking at very slow speed for ten minutes.
  Arms: Endurance exercise group
Other: Kinesiotaping — The participants will be asked to assume standing position then to flex back to reach its maximum point.
  * Two bands, 1 on each side of the lumbar spine, will be applied vertically from the lower posterior iliac crest region to the upper twelfth rib region, with inhibition technique.
  * The remaining 2 bands will be attached horizontally, with space correction technique.
  * All 4 bands will be placed to allow for 50% longitudinal stretching. The stretching directions for the vertical and horizontal applications were bottom-up and sideways, respectively.
  Arms: Kinesiotaping group

SUMMARY:
This study will be conducted to determine the effect of kinesiotaping versus endurance exercise on postmenopausal low back pain.

DETAILED DESCRIPTION:
Non-specific back pain is more frequent in women than men, mainly in postmenopausal women. High prevalence of hypovitaminosis D has been detected in postmenopausal women, and it is associated with decreased bone mass, sarcopenia, which can be related to back pain.

Postural control, can be defined as "the ability to maintain the body's center of gravity within the limits of stability as determined by the base of support , Differences in motor behavior between Low Back Pain (LBP) patients and healthy control subjects have been demonstrated in a variety of tasks, e.g. during walking and in response to several perturbations.

Published evidence indicates that LBP patients may have impaired control over trunk posture and movement, Dynamic controls is important in many functional tasks as it requires integration of appropriate levels of proprioception, range of motion, and strength. Endurance exercise is characterized by continues submaximal muscular contractions . It is an effective mean of maintaining or improving cardiovascular and musculoskeletal health, both of which are critical for preserving physiological functioning, independence and improving standing balance.

kinesiotape allows the joint to move through its full range of motion. It has also been reported to increase blood circulation and lymphatic drainage, which leads to a reduction of pain and stimulates large-fibre cutaneous mechanoreceptors that may inhibit proprioceptive impulses in the spinal column and decrease pain via an ascending pathway.

ELIGIBILITY:
Inclusion Criteria:

* A convenient sample of fifty postmenopausal women suffering from non-specific low back pain and postural instability was enrolled in this study.
* Praticipants were chosen healthy and medically stable.
* Their ages ranged from 50 - 60 years to be included in the study.
* Their body mass index (BMI) is not exceed 35 kg m2.
* All of them are diagnosed by the gynecologist.

Exclusion Criteria:

* They were excluded from the study if they had:
* Premature menopause or surgical menopause.
* Mental , neurological , vestibular , cardiovascular disorders, metabolic disease. -----
* Musculoskeletal disorders ( disc lesion , ankylosing spondylitis , rheumatoid arthritis , osteomalacia , spinal deformities, lumber vertebre fractures) .

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2025-01-16 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Pain level assessment: | 3 months
  Assessment of pain level for all participants will be measured before and after the treatment program by using the visual analogue scale (VAS) which is valid and reliable measure for pain intensity. It is a 10 cm horizontal line with two ends, 0 at one end which means no pain and 10 at the other end which means worst pain.

SECONDARY OUTCOMES:
Timed "Up and Go"Test (TUGT): | 3 months
  It will be used to evaluate postural balance for all participants in both groups before and after end of the treatment. it will be used to determine how many seconds the individual takes to perform the task of rising from a standard chair (seat approximately 46cm and arms 65cm high), walking 3 meters, turning around, returning to and sitting back on the chair. The participants will be instructed to perform at their usual speed and not enter into dialogues, They should have their usual footwear and if necessary a cane. Ten seconds to run the test was considered as a normal healthy adult performance; a period of 20 seconds is considered normal for frail elderly or disabled; however, a period above 20 seconds indicates the need to observe the level of functional impairment of the subject.
Unipodal stance test | 3 months
  It is a simple and good predictor of falls to evaluate the performance of the individual instructed to remain in single leg stance on each leg with eyes open or closed.
  The test starts with the legs parallel, maintaining a base of 10 cm away from the midline of each calcaneus, with the upper limbs hanging along the body. The subject is instructed to fix his gaze on a point that is at eye level and at a distance of one meter. Then, the examiner instructs the subject to take one foot from the ground, performing a hip flexion, and records the time during which the individual remains in position. The stay-in-position for more than 30 seconds indicates low risk of falling, whereas a time shorter than 5 sec shows a high risk of falls
Evaluation of core endurance | 3 months
  McGill's Core endurance tests will be used to evaluate core endurance for all participants in both groups before and after the end of the treatment. For the trunk anterior flexor test, participants sit with their backs flat against a wooden wedge angled at 60° with hands across their chest and their knees both flexed to a 90-degree angle as determined by a goniometer (Time recording is started when the wedge is moved back 10 cm and stopped when the trunk is deviated either forward or backward from the 60° angle

CONTACTS AND LOCATIONS:
Overall Officials: Hossam Hussien, Professor, Study Director — Al-Azhar University; Soheir El-kosery, Professor, Study Chair — Cairo University
Locations (1):
- Asmaa Mohamed Gaballah, Giza, Egypt